CLINICAL TRIAL: NCT02314975
Title: Intermittent Vibrational Force and Orthodontic Tooth Movement: a Randomised Controlled Trial
Brief Title: Intermittent Vibrational Force and Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/LO/0056
Record Dates: First submitted 2014-11-25; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Dental Crowding; Vibrational Force; Fixed Orthodontic Appliances
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AcceleDent vibrational device (Experimental): Fixed appliances with supplementary vibrational force
  Interventions: Device: AcceleDent vibrational device
- Sham AcceleDent device (Sham Comparator): Fixed appliances with supplementary sham device
  Interventions: Device: Sham AcceleDent device
- Fixed appliance only (Active Comparator): Fixed appliances only
  Interventions: Other: Fixed appliance only

INTERVENTIONS:
Device: AcceleDent vibrational device — Supplementary vibrational force with fixed appliances
  Arms: AcceleDent vibrational device
Device: Sham AcceleDent device — Supplementary sham-vibrational device with fixed appliances
  Arms: Sham AcceleDent device
Other: Fixed appliance only — Fixed appliance treatment only
  Arms: Fixed appliance only

SUMMARY:
The aim of this study is to compare the clinical efficiency of conventional fixed appliance orthodontic treatment with that supplemented by the daily application of cyclic forces to the dentition via a removable (AcceleDent) vibrational appliance. The primary outcome measure is rapidity of tooth alignment; whilst secondary outcome measures include pain and discomfort during treatment, rapidity of orthodontic space closure, changes in arch dimensions and root length.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from a sample of consecutive cases attending for routine fixed appliance orthodontic treatment with conventional pre-adjusted edgewise brackets that satisfy the following criteria: in the permanent dentition; a requirement for extraction of a premolar unit in each quadrant; incisor irregularity between 5-12 mm.

Exclusion Criteria:

* no medical contraindications; no craniofacial anomalies or cleft lip/palate;

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Orthodontic tooth movement (incisor alignment) | 2-12 months from start
  Irregularity (crowding) of the mandibular (lower) dental arch will be measured as total contact point displacement between the six canine and incisor teeth using digital calipers (150mm ISO 9001 electronic calliper, Tesa Technology, Renens, Switzerland; resolution ± 0.01mm) from stone dental casts. Initial crowding will be measured at T1 prior to the start of treatment. Irregularity will then be measured at T2 (at first archwire change) and the initial rate of orthodontic tooth movement calculated. Irregularity will then be measured at T3 (final alignment of the teeth) to calculate overall rate of alignment.

SECONDARY OUTCOMES:
Discomfort during initial orthodontic tooth movement | 1 week from start
  Subjects will fill out a questionnaire relating to their experiences of pain and discomfort during the first week of fixed appliance treatment. They will be asked to rate their pain on a 10-point visual analogue scale (no pain to extreme pain) at four time-points (4 hours; 24 hours; 3 days and 1 week) following placement of the appliance. They will also record the type and quantity of any analgesia taken during this time
Orthodontic space closure | 6-30 months from start
  Orthodontic space closure will be measured as the residual distance between canine and second premolar tooth using digital calipers from stone dental casts. This distance will be measured at each visit during space closure to calculate initial and overall rate of space closure.
Root resorption | 6-12 months from start
  Root length of the four lower incisor teeth will be measured from a long-cone periapical radiograph taken at the start of treatment (R1) using digital callipers. A second periapical radiograph of the lower incisors will be taken following tooth alignment (R2). The length of the crown from the tip to the cemento-enamel junction will also be measured at the start (C1) and end of alignment (C2). The X-ray enlargement factor will then be calculated as C1/C2, with apical root resorption = R1-R2 x (C1/C2)

REFERENCES:
- [Derived] DiBiase AT, Woodhouse NR, Papageorgiou SN, Johnson N, Slipper C, Grant J, Alsaleh M, Khaja Y, Cobourne MT. Effects of supplemental vibrational force on space closure, treatment duration, and occlusal outcome: A multicenter randomized clinical trial. Am J Orthod Dentofacial Orthop. 2018 Apr;153(4):469-480.e4. doi: 10.1016/j.ajodo.2017.10.021. PMID 29602338
- [Derived] DiBiase AT, Woodhouse NR, Papageorgiou SN, Johnson N, Slipper C, Grant J, Alsaleh M, Cobourne MT. Effect of supplemental vibrational force on orthodontically induced inflammatory root resorption: A multicenter randomized clinical trial. Am J Orthod Dentofacial Orthop. 2016 Dec;150(6):918-927. doi: 10.1016/j.ajodo.2016.06.025. PMID 27894540
- [Derived] Woodhouse NR, DiBiase AT, Johnson N, Slipper C, Grant J, Alsaleh M, Donaldson AN, Cobourne MT. Supplemental vibrational force during orthodontic alignment: a randomized trial. J Dent Res. 2015 May;94(5):682-9. doi: 10.1177/0022034515576195. Epub 2015 Mar 10. PMID 25758457